CLINICAL TRIAL: NCT03564054
Title: Multi-Center, Randomized Trial of Photodynamic Therapy Versus Argon Plasma Coagulation for Lung Cancer With Endobronchial Obstruction
Brief Title: Trial of Photodynamic Therapy Versus Argon Plasma Coagulation for Lung Cancer With Endobronchial Obstruction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual
Sponsor: University of Florida (Other)
Collaborators: Concordia Laboratories Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UF-THO-001; RGA030 (Other Grant/Funding Number: Concordia Laboratories, Inc.); UF-PDO-THO-1001 (Other: University of Florida Cancer Center); OCR17811 (Other: University of Florida)
Record Dates: First submitted 2018-06-08; First posted 2018-06-20 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: non small cell lung cancer; photodynamic therapy; argon plasma coagulation; endobronchial obstruction
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Photochemotherapy; Argon Plasma Coagulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Photodynamic Therapy (Experimental): Photodynamic therapy (PDT) uses activation of a photosensitizer by light of a specific wavelength to generate reactive oxygen species and singlet oxygen that causes direct cell damage and death, apoptosis, tumor vasculature damage and thrombosis, and inflammation leading to an immunological response.Following randomization, subjects will undergo treatment with either PDT or APC. Subjects will then have six additional study visits at 30, 45, 60, 90, and 180 days after their last PDT or APC treatment
  Interventions: Procedure: Photodynamic Therapy
- Argon Plasma Coagulation (Experimental): Argon plasma coagulation (APC) is a noncontact form of electrocautery. Following randomization, subjects will undergo treatment with either DPT or APC. Subjects will then have six additional study visits at 30, 45, 60, 90, and 180 days after their last PDT or APC treatment.
  Interventions: Procedure: Argon Plasma Coagulation

INTERVENTIONS:
Procedure: Photodynamic Therapy — Participants on this arm will be treated with photodynamic therapy. PDT is a two-stage process. The first stage of PDT is the intravenous injection of porfimer sodium (Photofrin) administered as a single slow intravenous injection over 3 to 5 minutes. The second stage involves the application of laser light to the tumor by bronchoscopy.
  Arms: Photodynamic Therapy
Procedure: Argon Plasma Coagulation — Participants on this arm will be treated with argon plasma coagulation. A flexible probe housing a wire delivers high-frequency, high-voltage electric current to a monopolar tungsten electrode present at the tip of the probe. Argon gas flows through the probe, and is charged or ionized to produce "plasma" as it flows around the tungsten electrode. Electric current flows through the plasma to the nearest tissue, and heat is produced as it passes through the tissue. Increased resistance created by coagulated tissue impairs the flow of electric current, and keeps the ablation depth to 1 to 2 mm.
  Arms: Argon Plasma Coagulation

SUMMARY:
The purpose of the study is to assess the efficacy of photodynamic therapy (PDT) in relieving airway obstruction in subjects with lung cancer compared to treatment with argon plasma coagulation (APC).

DETAILED DESCRIPTION:
This is a multi-center, randomized study that will compare the efficacy of photodynamic therapy (PDT) and argon plasma coagulation (APC) in the treatment of airway obstruction caused by non small cell lung cancer. Participants will be randomized in a 1:1 ratio to receive treatment with one of these two treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the subject and the ability for the subject to comply with all the study-related procedures.
* Subjects must have a biopsy proven for non-small cell lung cancer with obstructing or partially obstructing endobronchial tumor involving the main stem bronchus or bronchus intermedius, or lobar bronchus with or without extrabronchial tumor.
* Both males and females ≥ eighteen years of age
* Subject must demonstrate at least a 50% airway stenosis due to endobronchial tumor.
* Subject must demonstrate symptoms of cough, hemoptysis, dyspnea etc. attributable to partially or completely occluding endobronchial tumor.
* Subject is able to tolerate multiple bronchoscopies.
* Subjects who were previously treated with chemotherapy or radiotherapy are eligible for study entry. Such subjects must be at least 2 weeks post-radiotherapy and must have recovered from all acute toxicities associated with such treatment.
* A predicted life expectancy of at least 90 days.

Exclusion Criteria:

* Prior treatment of non-small cell carcinoma with PDT or with APC in the last 3 months.
* Subjects with tracheal lesions or carinal lesions that compromise both main stem bronchi.
* Subjects who have undergone pneumonectomy.
* Tumor involving or eroding into major blood vessels.
* Presence of a tracheoesophageal or bronchoesophageal fistula.
* Subjects receiving concurrent external beam radiation therapy.
* Radiation therapy within the previous two weeks.
* Inability to adhere to sunlight precautions.
* Severe hepatic impairment.
* Severe renal impairment.
* Porphyria or hypersensitivity to porphyrins.
* Subjects requiring supplemental O2 with a flow of greater than 3 lpm to keep resting oxygen saturations greater than 90%.
* History of any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy or that might affect the interpretation of the results of the study or that puts the subject at high risk for treatment complications, in the opinion of the treating physician.
* Prisoners or subjects who are involuntarily incarcerated.
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.
* Subjects demonstrating an inability to comply with the study and/or follow-up procedures.
* Females who are pregnant.
* Individuals who cannot provide consent themselves.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Treatment time until failure | 90 days
  Measure the time until treatment failure. Treatment failure is defined in this study as the occurrence of any of the following: failure to improve airway patency, airway-re-obstruction, need for additional airway intervention, and/or worsening symptoms at 90 days after the last PDT or APC treatment .

SECONDARY OUTCOMES:
Change in mean score of quality of life using the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire and Lung Cancer Module (EORTC QLQ-LC13) at 30, 90 and 180 days after the last PDT or APC | 30 days through 180 days
  QLQ-LC13 incorporates one multi-item scale to assess dyspnoea, and a series of single items assessing pain, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and haemoptysis. All of the scales and single-item measures range in score from 0 to 100. A high score for the scales and single items represents a high level of symptomatology or problems.
Need for additional bronchoscopic therapies for either endobronchial obstruction at the treated site or for recurrent obstruction with no additional therapies offered at 30, 90, and 180 days following the last PDT or APC treatment | 30 days through 180 days
  This will be assessed as Yes/No at each of the time points as to whether additional bronchoscopic therapies are needed, in the opinion of the treating investigator
Median survival time | 6 months
  The median survival time for each treatment cohort will be estimated in days after the last PDT or APC treatment using a Kaplan-Meier survival curve
Percent reduction in airway obstruction as measured by bronchoscopy at 30 and 90 days after the last PDT or APC treatment | 30 days through 90 days
  Percent reduction in airway obstruction will be calculated with the formula: [(baseline obstruction percentage - residual obstruction percentage)/baseline obstruction percentage x 100%].
Resolution of atelectasis, if present, at 30, 45, 60, 75, 90, and 180 days after the last PDT or APC treatment | 30 days through 180 days
  This will be assessed by examining subject chest x-rays and/or chest CT scans at each of these time points for the presence or absence of atelectasis.
Resolution of post-obstructive pneumonia, if present, at 30, 45, 60, 75, 90, and 180 days after the last PDT or APC treatment | 30 days through 180 days
  This will be assessed by examining subject chest x-rays and/or chest CT scan for the presence or absence of post-obstructive pneumonia, as well as the physical examination of subjects for post-obstructive pneumonia symptoms (such as fever, pleuritic chest pain, and productive cough) at each of these time points.
Change in dyspnea (as measured by the transitional dyspnea index (TDI), using the score obtained from the Baseline Dyspnea Index (BDI) as the baseline comparator) at 30, 60, 90, and 180 days after the last PDT or APC treatment | 30 days through 180 days
  The Baseline Dyspnea Index measures the severity of dyspnea at baseline using the sum of the scores for three items that assess functional impairment and magnitude of effort required for daily activities. Total possible score ranges from 0 to 12. A lower total score indicates more severe dyspnea. The Transitional Dyspnea Index evaluates change in dyspnea as compared to the score obtained by the Baseline Dyspnea Index using a scale of -9 to +9. A negative score (-1 to -9) indicates worsening dyspnea as compared to baseline, a positive score (+1 to +9) indicates improvement in dyspnea as compared to baseline, and a score of 0 indicates no change in dyspnea as compared to baseline.
Change in hemoptysis, if present, at 30, 45, 60, 75, 90, and 180 days after the last PDT or APC treatment using categorical measures (worsened, unchanged, improved, resolved) | 30 days through 180 days
Change in cough, if present, at 30, 45, 60, 75, 90, and 180 days after the last PDT or APC treatment using categorical measures (worsened, unchanged, improved, resolved) | 30 days through 180 days
Change in Karnofsky performance status, if present, at 30, 60, 90, and 180 days after the last PDT or APC treatment using categorical measures (worsened, unchanged, improved, resolved). | 30 days through 180 days
Proportion of patients experiencing treatment failure at 90 days | 90 days
  Treatment failure is defined as failure to improve airway patency, airway re-obstruction, need for additional airway intervention and/or worsening symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jantz, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States